CLINICAL TRIAL: NCT00423878
Title: Clinical Management of Metabolic Problems in Patients With Schizophrenia
Brief Title: Comparison of Antipsychotics for Metabolic Problems in Schizophrenia or Schizoaffective Disorder
Acronym: CAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STROUP06STN0; DSIR AT-AP (Other: National Institute of Mental Health)
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Olanzapine; Quetiapine Fumarate; Aripiprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will switch to aripiprazole with a cross-titration from the current antipsychotic over 3-4 weeks. Allowed final dosage range for aripiprazole was 5-30 mg/day
  Interventions: Drug: Aripiprazole
- 2 (Active Comparator): Participants will continue with their current antipsychotic treatment, either olanzapine 5-20 mg/day, quetiapine 200-1200 mg/day, or risperidone 1-16 mg/day.
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Quetiapine

INTERVENTIONS:
Drug: Risperidone — Continued treatment with the medication risperidone for schizophrenia for up to 6 months in study
  Other Names: Risperdal
  Arms: 2
Drug: Olanzapine — Continued treatment with the medication olanzapine for schizophrenia for up to 6 months in study
  Other Names: Zyprexa
  Arms: 2
Drug: Quetiapine — Continued treatment with the medication quetiapine for schizophrenia for up to 6 months in study
  Other Names: Seroquel
  Arms: 2
Drug: Aripiprazole — Switching medication to aripiprazole for schizophrenia for up to 6 months in study
  Other Names: Abilify
  Arms: 1

SUMMARY:
The study will compare the effectiveness of antipsychotic medications for patients with schizophrenia or schizoaffective disorder for whom a medication change may be indicated because of an increased risk of cardiovascular disease.

DETAILED DESCRIPTION:
Metabolic abnormalities associated with cardiovascular morbidity and premature mortality are more common in patients with schizophrenia than in matched controls. Although there is some evidence that patients with schizophrenia have intrinsic abnormalities in lipid and carbohydrate metabolism, some antipsychotics (i.e., clozapine, olanzapine, quetiapine, and risperidone) are associated with increased rates of metabolic abnormalities that predispose patients to cardiovascular disease.

This is an investigator-initiated clinical trial that will be conducted at 30 research sites that are a part of the NIMH Schizophrenia Trials Network.

The aims of the study are to (1) determine the relative effects of switching to aripiprazole, versus continued treatment with olanzapine, quetiapine, or risperidone, on metabolic parameters associated with cardiovascular disease, and (2) to determine the effects of switching to aripiprazole versus continued treatment with olanzapine, quetiapine, or risperidone on the clinical stability of schizophrenic illness.

This study design is a multi-site, single-blind (rater) randomized controlled trial of 300 patients with schizophrenia or schizoaffective disorder comparing treatment with the following medications: olanzapine, quetiapine, risperidone, and aripiprazole. The study will enroll patients with schizophrenia or schizoaffective disorder for whom a medication change may be indicated because of an increased risk of cardiovascular disease in spite of adequate control of symptoms on their current antipsychotic medication. Patients who are taking olanzapine, quetiapine, or risperidone and who have a body-mass index (BMI) greater than or equal to 27 and non-HDL cholesterol greater than or equal to 130 mg/dl will be eligible (if non-HDL is between 130-139mg/dL, LDL cholesterol must be greater than 100mg/dL). All treatments will be open label. Raters will be blinded to treatment assignment. Patients will be followed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia or schizoaffective disorder
* Currently treated with olanzapine, quetiapine or risperidone
* BMI greater than or equal to 27
* Non-HDL cholesterol greater than or equal to 130 mg/dL (if non-HDL cholesterol is between 130 - 139 mg/dL, then LDL cholesterol must be greater than 100 mg/dL).

Exclusion Criteria:

* Diabetes (FBS greater than or equal to 126) or treatment with oral hypoglycemic drug or insulin
* Non-HDL cholesterol greater than 300 mg/dL
* Serum triglycerides greater than 500 mg/dL
* Patients in the first episode of schizophrenia or schizoaffective disorder
* Known hypersensitivity to aripiprazole
* On weight loss medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Scott Stroup, MD, MPH, Principal Investigator — Columbia University; Joseph P. McEvoy, MD, Study Director — Duke University
Locations (28):
- United States (28):
  - SHANTI Clinical Trials, Colton, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Mental Health Advocates, Boca Raton, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Clinical Research Institute, Wichita, Kansas
  - Lousiana State University Health Sciences Center, Shreveport, Louisiana
  - Clinical Insights, Glen Burnie, Maryland
  - Freedom Trail Clinic, Boston, Massachusetts
  - John C Corrigan Community Mental Health Center, Fall River, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - Research Foundation for Mental Hygiene, New York, New York
  - University of Rochester, Rochester, New York
  - John Umstead Hospital/Duke University, Butner, North Carolina
  - The University of North Carolina, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Philadelphia VA Medical Center-116A, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Stroup TS, McEvoy JP, Ring KD, Hamer RH, LaVange LM, Swartz MS, Rosenheck RA, Perkins DO, Nussbaum AM, Lieberman JA; Schizophrenia Trials Network. A randomized trial examining the effectiveness of switching from olanzapine, quetiapine, or risperidone to aripiprazole to reduce metabolic risk: comparison of antipsychotics for metabolic problems (CAMP). Am J Psychiatry. 2011 Sep;168(9):947-56. doi: 10.1176/appi.ajp.2011.10111609. Epub 2011 Jul 18. PMID 21768610

RESULTS

PARTICIPANT FLOW:
Groups:
- Switch Group: Participants will switch to aripiprazole with a cross-titration from the current antipsychotic over 3-4 weeks. Allowed final dosage range for aripiprazole was 5-30 mg/day.
- Stay Group: Participants will continue with their current antipsychotic treatment, either olanzapine 5-20 mg/day, quetiapine 200-1200 mg/day, or risperidone 1-16 mg/day.
Period: Overall Study
Arm/Group | Switch Group | Stay Group
Started | 109 | 106
Completed | 89 | 98
Not Completed | 20 | 8

BASELINE CHARACTERISTICS:
Groups:
- Switch Group: Participants will switch to aripiprazole.
- Stay Group: Participants will continue treatment with olanzapine, quetiapine, or risperidone.
- Total: Total of all reporting groups
Arm/Group | Switch Group | Stay Group | Total
Number analyzed (Participants) | 109 | 106 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 106 | 215
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.7) | 42 (10.5) | 41 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 37 | 78
  Male | 68 | 69 | 137
Region of Enrollment [Number; unit: participants]
  United States | 109 | 106 | 215
non-HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 169 (31.9) | 176 (33.5) | 173 (32.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-HDL Cholesterol Level for Patients Assigned to Stay and Patients Assigned to Switch Over 24 Weeks
Description: Change in non-HDL cholesterol measured at baseline and every 4 weeks for 24 weeks. The efficacy analysis corresponded to a comparison of change in non-HDL cholesterol from baseline to 24 weeks between treatment groups (stay versus switch). Repeated measurements mixed effects linear models were fit for the primary analysis.
Time Frame: 24 weeks
Population: The primary efficacy analysis was conducted on the efficacy evaluable population, defined as all patients randomly assigned to a study group who received at least one dose of study medication and completed at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: mg/dL non-HDL cholesterol
Arm/Group | Switch Group | Stay Group
Number analyzed (Participants) | 89 | 98
mg/dL non-HDL cholesterol | -20.2 (2.87) | -10.8 (2.57)

2. Secondary Outcome: Efficacy Failure, Defined as Psychiatric Hospitalization, a 25 Percent Increase From Baseline on the Positive and Negative Syndrome Scale or Substantial Clinical Deterioration on the Clinical Global Impressions-Change (CGI-C)
Time Frame: Measured at Month 6
Population: 2 participants who never took assigned study medication were excluded.
Measure: Number; unit: participants
Arm/Group | Switch Group | Stay Group
Number analyzed (Participants) | 107 | 106
participants | 22 | 18

ADVERSE EVENTS:
Description: Two participants randomized to switch to aripiprazole withdrew from the study before taking the study medication.
Arm/Group | Switch Group | Stay Group
Serious Adverse Events (participants affected / at risk) | 18/107 | 9/106
Other Adverse Events (participants affected / at risk) | 77/107 | 77/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch Group (N=107) | Stay Group (N=106)
Exacerbation of schizophrenia (Psychiatric disorders) | 9 (11) | 3 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Slurred speech/sedation (General disorders) | 1 (2) | 0 (0)
Suicidality (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accidental overdose (General disorders) | 1 (1) | 1 (1)
Neuropathic pain (Nervous system disorders) | 1 (1) | 0 (0)
Victim of gunshot wound (General disorders) | 1 (1) | 0 (0)
(General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch Group (N=107) | Stay Group (N=106)
Insomnia (Psychiatric disorders) | 44 (44) | 29 (29)
Sleepiness (Psychiatric disorders) | 27 (27) | 35 (35)
Dry mouth (Gastrointestinal disorders) | 24 (24) | 36 (36)
Akathisia/activation (Nervous system disorders) | 29 (29) | 26 (26)
Problems with sex drive (Endocrine disorders) | 24 (24) | 26 (26)
Increased appetite (General disorders) | 18 (18) | 26 (26)
Weight gain (General disorders) | 20 (20) | 21 (21)
Constipation (Gastrointestinal disorders) | 20 (20) | 20 (20)
Akinesia (Nervous system disorders) | 14 (14) | 25 (25)
Problems with sexual orgasm (Endocrine disorders) | 20 (20) | 19 (19)
Problems with sexual arousal (Endocrine disorders) | 20 (20) | 18 (18)
Hypersomnia (General disorders) | 16 (16) | 21 (21)
Orthostatic faintness (General disorders) | 19 (19) | 18 (18)
Nausea (Gastrointestinal disorders) | 12 (12) | 18 (18)
Incontinence/nocturia (Renal and urinary disorders) | 9 (9) | 13 (13)
Skin rash (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (12)
Menstrual irregularities (Endocrine disorders) | 10 (10) | 6 (6)
Sialorrhea (General disorders) | 8 (8) | 7 (7)
Urinary hesistancy (Renal and urinary disorders) | 5 (5) | 4 (4)
Gynecomastia/galactorrhea (Endocrine disorders) | 2 (2) | 4 (4)

LIMITATIONS AND CAVEATS:
Open-label treatment is a limitation of this study, particularly for outcomes not measured in the laboratory but instead subject to clinical judgment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No